CLINICAL TRIAL: NCT01041482
Title: A Multi-Center, Non-Controlled Clinical Study of Sorafenib Adjuvant Therapy in Locally Advanced Renal-Cell Carcinoma After Radical Nephrectomy
Brief Title: A Multi-Center, Non-Controlled Clinical Study of Sorafenib Adjuvant Therapy in Advanced Renal-Cell Carcinoma
Acronym: AGuo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing University of Chinese Medicine (Other); China Medical University, China (Other); Peking Union Medical College Hospital (Other); Tianjin Medical University (Other); Shanghai Jiao Tong University School of Medicine (Other); Changhai Hospital (Other); Zhejiang University (Other); Fudan University (Other); Jiangsu Province Centers for Disease Control and Prevention (Network); Central South University (Other); Sichuan University (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bay 43-9006
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2008-08

CONDITIONS: Renal Cell Carcinoma
Keywords: sorafenib; renal cell carcinoma; disease free survival; Hand food skin reaction
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib (Experimental): To study the efficacy of Sorafenib as an adjuvant therapy for reducing recurrence rate in locally advanced renal-cell carcinoma (RCC) after radical nephrectomy.
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — sorafenib 400mg twice daily

SUMMARY:
A one-arm,open,multi-center study, to evaluate sorafenib (400mg twice daily ) as a adjuvant to prevent recurrence of RCC(renal cell carcinoma) patients after radical nephrectomy with a high-risk of recurring. To observe disease-free survival and the survival rate in 3 years,5 years.

The purpose of this study is:

* To study the efficacy of Sorafenib as an adjuvant therapy for reducing recurrence rate in locally advanced renal-cell carcinoma (RCC) after radical nephrectomy.
* To observe the incidence of hand-foot skin reaction (HFSR) after the Urea (10% or 5%) based cream intervention treatment.

The primary end point is the disease-free survival(DFS).The secondary end point is overall survival(OS),the drug safety and tolerance, the occurrence of hand foot skin reaction(HFSR) at the week of 3,6,12,the skin toxicity(not include HFSR) higher than CTCAE(Common Terminology Criteria for Adverse Events) Grade 2 at the 12th week, the incidence of HFSR after the Urea (10% or 5%) based cream intervention treatment.

DETAILED DESCRIPTION:
A one-arm, open, multi-center study, to evaluate sorafenib (400mg twice daily) as a adjuvant to prevent recurrence of RCC(renal cell carcinoma) patients after radical nephrectomy with a high-risk of recurring. To observe disease-free survival and the survival rate in 3 years, and 5 years. To observe the incidence of hand-foot skin reaction (HFSR) after the Urea (10% or 5%) based cream intervention treatment. 140 subjects are prospected to enter the trial.

The sorafenib adjuvant therapy is unremitting with a time of 12 months. For a convenient record, every 6 weeks is regarded as a single observational cycle. The end-point are recurrence, not being tolerant to the toxicity, need to stop the intervening study or withdrawing the informed consent. It is necessary to evaluate the efficacy and safety every 6 weeks. At the screening stage and every 12 weeks imaging review are performed such as abdominal and chest CT or MRI, the imaging methods of a single subject should be in uniformity during the trial.

The post-treatment evaluation are performed 30 days after the last usage of the adjuvant in order to collect all the adverse events (AE) and the survival rates of all the subjects. The agent-relevant AE (known or unknown) should be reported to the drug safety institution, the patients should be visited until the events solved, except the events can not be solved for the subjects' underlying diseases.

ELIGIBILITY:
Inclusion Criteria:

Preoperative Criteria

* Renal local advanced renal cell carcinoma and be suitable to radical nephrectomy.
* Tumor >=7cm, the lymph nodes in metastasis can be resectable, the renal vein or inferior caval vein with metastatic thrombus can be resectable also, clinical staging>=T2anyNMo.
* Resectable tumor with multiple-lesion in ipsolateral kidney Enrolment Criteria
* No distant metastasis.
* Not undergoing any adjuvant or systematic anti-tumor therapy, such as chemotherapy, biotherapy or radiotherapy.
* After the nephrectomy 4-12 weeks and should be recovery in the postoperative complications.
* ECOG scores 0-1.
* Referring to the Scoring Algorithm to Predict Metastasis after Radical Nephrectomy in Patients with clear cell renal cell carcinoma, all the patients score higher than 6. Metastatic lymph node with clinical diagnosis have been resected, all the resected specimen edge be negative in pathological detection.

The pathological diagnosis of renal cell carcinoma:

* No remnant tumor with postoperative imaging screening with CT or MRI.
* The liver and renal function, hemocytogenesis function meet the below criteria within the 4 weeks before the enrollment.

  * Granulocytes count >1500/mm3
  * Blood platelet >100000/mm3
  * Creatinine<2 times of the upper of the reference value
  * Total bilirubin<1.5 times of the upper of the reference value
  * Alanine aminotransferase/aspartate aminotransferase<2.5 times of the upper of the reference value
  * The informed consent has been endorsed.

Exclusion Criteria:

* Other coincident carcinoma, but not including carcinoma in situ of cervix and basal cell epithelioma after radical therapy and bladder carcinoma superficially(Ta,Tis,T1) or carcinoma having been cured 3 years ago.
* Cardiac dysrhythmia need agent intervention(not including β-receptor inhibitive or digoxin treatment), coronary heart disease, myocardial infarction occurred in the later 6 months, heart failure assessment higher than NYHA II
* Seriously active infection with bacteria or fungus
* HIV infection or HBV/HCV infection with IFN-a intervention.
* Dysfunction in blood coagulation.
* Epilepsia with drug treatment.
* Those cannot take tablets orally.
* Allogeneic organ transplantation.
* Drug abuse or concomitant conditions such as psychologically or socially factors which may intervene the assessment.
* Hypersensitiveness to the studying adjuvant or the trial-relevant drugs.
* Pregnancy or lactation, pregnancy test must be negative within the 14 days before the trial beginning, either females or males must be contraceptive during the trial.
* The following concomitant therapeutics must be excluded:

  * Anti-tumor agents, immunological or hormonal therapy
  * Radiotherapy
  * Biological therapeutics such as G-CSF or GM-CSF
  * Autologous bone marrow transplantation or stem cell treatment
  * The other trial medicine therapeutics
  * Bevacizumab treatment or other agents effected in VEGF or VEGF-receptor, such as inhibitive in Raf or MEK

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
disease free survival | November 2008-November 2013

SECONDARY OUTCOMES:
overall survival | November 2008-November 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Jianhui Ma, Beijing, Beijing Municipality, China